CLINICAL TRIAL: NCT06614569
Title: Long-Term Follow-Up of A Two-Stage Dose-Escalation Study to Evaluate the Safety and Efficacy of Bilateral Intraparenchymal Thalamic and Intracisternal/Intrathecal Admin of AXO-AAV-GM2 in Tay-Sachs or Sandhoff Disease
Brief Title: Long-Term Follow-Up of Subjects Treated With AXO-AAV-GM2 for Tay-Sachs or Sandhoff Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Terence Flotte (Other)
Responsible Party: Sponsor-Investigator, Terence Flotte, Professor and Dean, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: STUDY00001894
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: GM2 Gangliosidosis; Tay Sachs Disease; Sandhoff Disease
MeSH Terms: conditions — Gangliosidoses, GM2; Tay-Sachs Disease; Sandhoff Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — May possibly retain frozen blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects previously treated with AXO-AAV-GM2 gene therapy for Tay-Sachs or Sandhoff Disease: All subjects have previously received gene therapy and will be followed for the collection of clinical information, especially pertaining to de novo cancer, neurologic, rheumatologic, and hematologic/immunologic disorders following AAV gene therapy.
  Interventions: Drug: AXO-AAV-GM2

INTERVENTIONS:
Drug: AXO-AAV-GM2 — Participants who received AXO-AAV-GM2 will be tracked in long term follow up

SUMMARY:
This study is to continue Long-Term Follow-Up of Patients who were previously treated with AXO-AAV-GM2 Gene Therapy as treatment for Tay-Sachs or Sandhoff Disease to follow the subjects through 5 years after their initial gene therapy treatment.

DETAILED DESCRIPTION:
Subjects will be contacted bi-annually for a total of five years following the administration of AXO-AAV-GM2 for the collection of clinical information, especially pertaining to de novo cancer, neurologic, rheumatologic, and hematologic/immunologic disorders. This will be done to comply with FDA Recommendations and NIH Guidelines for long-term follow-up for research involving gene therapy with AAV Vectors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously enrolled in the study "A Two-Stage Dose-Escalation Study to Evaluate the Safety and Efficacy of Bilateral Intraparenchymal thalamic and intracisternal/Intrathecal Admin of AXO-AAV-GM2 in Tay-Sachs or Sandhoff Disease."

Exclusion Criteria:

* Subjects who were not previously enrolled under the initial protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Tay-Sachs or Sandhoff Disease who were previously treated with AXO-AAV-GM2
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Long term Safety of AXO-AAV-GM2 | Every 6 months, up to five years
  Participants will be monitored for adverse events, including delayed adverse events, as a result of AXO-AAV-GM2 including de novo cancer, neurologic, rheumatologic, and hematologic/immunologic disorders.

SECONDARY OUTCOMES:
Long term Impact of AXO-AAV-GM2 | Every 6 months, up to five years
  Participants will be monitored for the impact of treatment with AXO-AAV-GM2 on the expected natural history of their condition in the domains of neurocognitive adaptive, developmental, neurological and motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Flotte, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eichler F, Cataltepe OI, Daci R, Puri AS, Taghian T, Jiang X, Shazeeb MS, Kuhn A, Hader A, Celik H, Vardar Z, Lewis CJ, Artinian R, Nagy A, Vachha B, Thompson R, Gallagher T, Bateman S, Parzych J, Spanakis SG, Vaughn TA, Pier K, De Boever E, Abbott MA, D Ambrosio E, Kokoski D, Blackwood M, Drummond E, Ratai EM, Townsend EL, McLaughlin H, Tifft CJ, Keeler AM, Sena-Esteves M, Gray-Edwards HL, Flotte TR. Dual-vector rAAVrh8 gene therapy for GM2 gangliosidosis: a phase 1/2 trial. Nat Med. 2025 Sep;31(9):2927-2935. doi: 10.1038/s41591-025-03822-4. Epub 2025 Aug 15. PMID 40817303